CLINICAL TRIAL: NCT00577915
Title: Breast MRI Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-037
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Suspicion of, or Known Breast Cancer
Keywords: Breast cancer; MRI spectroscopy; Diagnostic radiology
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Breast MR Spectroscopy (Experimental): Conventional images will be taken with standard pulse sequences. These images will be used for the diagnostic examination for which the patient will have been scheduled. Following the diagnostic study, a pulse sequence designed to obtain spectroscopy data will be used.This will be used on the existing magnets 1.5T and 3T. Memorial Sloan-Kettering Cancer Center has 1.5T and 3T magnets. The patient will have only one injection of contrast (gadolinium-DTPA) for the initial diagnostic study. No additional contrast will be administered. The additional sequence should take about 10 minutes, depending on breast size.
  Interventions: Other: Radiology/MRI scan

INTERVENTIONS:
Other: Radiology/MRI scan — MRI spectroscopy

SUMMARY:
The purpose of this study is to provide physicians with additional information not available with standard imaging methods for breast disease.

As part of the MRI examination ordered by your physician, a new method of analyzing the images or pictures will be used. This new method is called spectroscopy and is used routinely on other parts of the body such as the prostate and brain. Pictures produced with this sequence may look slightly different than the regular MRI pictures. Using spectroscopy data, it may be possible to distinguish benign conditions of the breast from malignant tumors and provide more precise information than can be obtained with regular MRI.

DETAILED DESCRIPTION:
Our aim is to perform MR Spectroscopy (MRS) on 150 evaluable patients at the end of their routine breast MRI examination using a software package from General Electric Medical Systems Milwaukee, WI). This will add time to the routine examination but will not involve additional injections of contrast. We will analyze the spectroscopic data to determine if benign lesions can be reliably differentiated from malignant ones.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for diagnostic breast MRI examination or interventional procedure for a known or suspected breast lesion

Exclusion Criteria:

* Patients who would be normally excluded from undergoing an MRI examination:

  * Patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To determine if spectroscopy of the breast can be performed and can be functional in a clinical environment. | 12 months

SECONDARY OUTCOMES:
To determine if the data obtained can be reliably analyzed and useful to the final interpretation of the breast MRI examination. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Brennan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org